CLINICAL TRIAL: NCT00389675
Title: A Double-Blind, Active-Controlled, Long-Term Safety Extension Study of Optimized Doses of Darusentan in Subjects With Resistant Hypertension Despite Receiving Combination Therapy With Three or More Antihypertensive Drugs, Including a Diuretic, as Compared to Guanfacine (Protocol DAR-312-E)
Brief Title: DORADO-AC-EX - A Long-Term Safety Extension Study to the Phase 3 DORADOC-AC Study (Protocol DAR-312) of Darusentan in Resistant Hypertension
Acronym: Darusentan
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study DAR-312 did not meet its primary co-endpoints.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol DAR-312-E
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — darusentan; Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darusentan (Experimental): Darusentan capsules titrated to an optimal dose of 50 mg, 100 mg, or 300 mg administered orally once daily
  Interventions: Drug: Darusentan
- Guanfacine (Active Comparator): Guanfacine 1 mg capsules administered orally once daily
  Interventions: Drug: Guanfacine

INTERVENTIONS:
Drug: Darusentan — Darusentan capsules at a dose of 50, 100, or 300 mg administered orally once daily
  Other Names: LU 135252
  Arms: Darusentan
Drug: Guanfacine — Guanfacine 1 mg capsules administered orally once daily
  Arms: Guanfacine

SUMMARY:
This is a double-blind, active-controlled, long-term study of a new experimental drug called darusentan. Darusentan in not currently approved by the United States Food and Drug Administration (FDA), which means that a doctor cannot prescribe this drug. The purpose of this study is to evaluate the long-term safety of darusentan (optimized dose) as compared to an active control, administered orally.

ELIGIBILITY:
SELECTED INCLUSION CRITERIA:

1. Subjects must be competent to provide written informed consent;
2. Subjects must have completed the Maintenance Period of the DAR-312 study.

SELECTED EXCLUSION CRITERIA:

1. Subjects who discontinue treatment with study drug prior to the end of the Maintenance Period in DAR-312 due to a study drug-related AE;
2. Subjects who experience a study drug-related serious adverse event (SAE) during the DAR-312 study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean 24-hour systolic and diastolic ambulatory blood pressure | Baseline to Week 14
Percentage of subjects who reach systolic blood pressure goal | Week 14
Change from baseline in estimated glomerular filtration rate (eGFR) | Baseline to Week 14

SECONDARY OUTCOMES:
Change from baseline in trough sitting systolic and diastolic blood pressures | Baseline to Week 14

CONTACTS AND LOCATIONS:
Locations (99):
- United States (85):
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - The Heart Center, PC, Huntsville, Alabama
  - Mulberry Medical Associates, PC, Montgomery, Alabama
  - Arizona Center for Clinical Research, Glendale, Arizona
  - Cardiovascular Consultants, Ltd., Glendale, Arizona
  - Lovelace Scientific Resource, Inc., Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Southwest Heart, Tucson, Arizona
  - HealthFirst Physicians of AR, PA dba Convenient Care Clinic, Hot Springs, Arkansas
  - NEA Clinical, Jonesboro, Arkansas
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Medical Investigators, Inc., Little Rock, Arkansas
  - Highgrove Medical Center, Bakersfield, California
  - Central Cardiology Medical Clinic, Bakersfield, California
  - Impact Clinical Trials, Beverly Hills, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Pacific Heart Institute, Santa Monica, California
  - Los angeles biomedical research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Doctors Medical center of Walton County, DeFuniak Springs, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Maxine Hamilton, MD, PA, Fort Lauderdale, Florida
  - St John's Center for Clinical Research, Jacksonville, Florida
  - Private Practice of Dr. Bridget Bellingar, Largo, Florida
  - A + Research Inc., Miami, Florida
  - AppleMed Research, Inc., Miami, Florida
  - Internal Medicine Associates of South Florida, North Miami Beach, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Nothwest Florida Heart Group, PA-Research Dept, Pensacola, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Suncoast Cardiovascular Research, Inc, St. Petersburg, Florida
  - Tampa Bay Nephrology Associates, PL, Tampa, Florida
  - Orlando Rangel, MD, PA, Tampa, Florida
  - AMR Research Associates, LLC, Bogart, Georgia
  - Atlanta Vascular Research Foundation, Tucker, Georgia
  - Consultants in Cardiovascular Med (CIS), Melrose Park, Illinois
  - Illinois Heart & Lunch Research Center, Normal, Illinois
  - Methodist Medical Center-Heart, Lung & Vascular Institute, Peoria, Illinois
  - Medical consultants, PC, Muncie, Indiana
  - University Medical Associates, Louisville, Kentucky
  - Dr. Jeffrey Chen, Lafayette, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Maine Research Associates, Auburn, Maine
  - PrimeCare Internal Medicine, Biddeford, Maine
  - Great Lakes Heart Center of Alpena, Alpena, Michigan
  - Internal Medicine of Northern Michigan, Petoskey, Michigan
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Central Minnesota Heart Center at St. Cloud Hospital, Saint Cloud, Minnesota
  - St. Paul Cardiology, Saint Paul, Minnesota
  - Glacier View Cardiology, PC, Kalispell, Montana
  - Impact Clinical Trials, Las Vegas, Nevada
  - NJ Heart, Linden, New Jersey
  - New Jersey Physicians, Passaic, New Jersey
  - Lifeline Research Institute, Brooklyn, New York
  - Metrolina Internal Medicine, PA, Charlotte, North Carolina
  - Heart Care Center of Charlotte, Charlotte, North Carolina
  - Physicians East, PA, Winterville, North Carolina
  - Plaza Medical Group, PC, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, LLC, Tulsa, Oklahoma
  - Integrated Medical Research PC, Ashland, Oregon
  - Blackstone Cardiology Associates, Pawtucket, Rhode Island
  - Charleston Cardiology, Charleston, South Carolina
  - Paris View Family Practice, Greenville, South Carolina
  - Internal Medicine of Greer, Greer, South Carolina
  - Scenic City Research, Cleveland, Tennessee
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Cardiovascular Research Inst. of Dallas, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Sergio F Rovner, MD, El Paso, Texas
  - Salim Gopalani, MD, PA, Houston, Texas
  - Humayum Mirza, MD, PA, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Houston Clinical Research Assoc., Houston, Texas
  - Innovative Research of West Florida, Hurst, Texas
  - North Texas Medical Research, Plano, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Fletcher Allen Health Care/University of Vermont, Burlington, Vermont
  - Kamlesh N Dave Cardiology, Hopewell, Virginia
  - WVU Physicicans of Charleston, Charleston, West Virginia
  - Alpha Medical Research, LLC, Madison, Wisconsin
  - Executive Health and Research Associates, Madison, Wisconsin
- Argentina (11):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca
  - Consultorios Medicos Privados S.A., Buenos Aires
  - Policlinica Bancaria "9 de Julio", Buenos Aires
  - Diabaid (Instituto de Asistencia Integral en Diabetes), Ciudad de Buenos Aires
  - MD Investigaciones, Ciudad de Buenos Aires
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Framingham Centro Medico, La Plata
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas de Quilmes, Quilmes
  - Instituto de Investigaciones Clinicas, Rosario
  - Centro de Investigaciones clincas de Litoral, Santa Fe
- Australia (2):
  - Flinders Medical Centre, Bedford
  - Royal Perth Hospital, Perth
- Private Practice of Dr. Herwig Van Aerde, Rio de Janeiro, Brazil

REFERENCES:
- See also: Related Info — http://www.gilead.com